CLINICAL TRIAL: NCT06930417
Title: Characterization and Natural History of Williams Syndrome and Other Chromosome 7q11.23 Variants
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Dasha Fleyshman, Research Program Manager, University of Pennsylvania
Other Study IDs: 851719; 23-020775 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2025-03-17; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Williams Beuren Syndrome; Williams Syndrome; Williams Beuren Region Duplication; Dup7
Keywords: williams syndrome; Dup7; svas; 7q11.23; autism
MeSH Terms: conditions — Williams Syndrome; Aortic Stenosis, Supravalvular; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (including PBMCs, plasma and serum); Post-surgery residual tissue; DNA (extracted from either blood cells or saliva)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational natural history study is to better characterize development, transition to adulthood, health and behavior of individuals diagnosed with Williams syndrome (WS) or carrying other variants of 7q11.23 chromosome and to build a DNA and tissue biobank with samples donated by affected individuals. The study has multiple arms focused on different aspects of WS. Participants with genetic diagnosis of WS or other variants of 7q11.23 and their family members are eligible to participate. Study participants may participate in one or multiple arms of the study:

1. Natural History Genotype-Phenotype Study to test the hypothesis that health, behavior, and developmental variability observed in WS is determined by genetic factors and to characterize those genetic changes. Participants of all ages are eligible to participate. Either a blood or saliva sample is required for participation.
2. Biobank: the research team is building a biobank enabling the development of new laboratory tools and models to study WS and test new treatment approaches. A blood sample is required for participation. Participants of all ages are eligible to participate.
3. Development arm of the study aims to delineate the development of language, cognition, personality, literacy and mathematics skills, and adaptive behavior from very early childhood through adulthood in individuals who have WS or Dup7. The purpose of this study also includes determining the predictors of specific aspects of development (e.g., word reading ability, language ability, spatial ability) for individuals with WS or Dup7. Affected individuals of all ages are eligible to participate.
4. Transition to Adulthood study aims to understand how young adults with WS make a successful transition out of high school into adulthood and to help them in this journey by providing a comprehensive psychosocial transition coupled with a medical transition plan. Individuals ages 14-25 years old are eligible to participate. Study requires three in person visits.

ELIGIBILITY:
Inclusion Criteria:

* clinical and/or molecular diagnosis of Williams syndrome (WS)
* biological parents or siblings of individuals diagnosed with WS
* molecular diagnosis of 7q11.23 duplication syndrome (Dup7)
* molecular diagnosis of another abnormality in the 7q11.23 region

Exclusion Criteria:

- No diagnosis of abnormalities in the 7q11.23 region, while not being a biological relative of affected individuals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a clinical and/or molecular diagnosis of Williams Syndrome, 7q11.23 duplication syndrome, or another abnormality in the 7q11.23 region and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2040-10-21 (Estimated); Study Completion 2045-10-21 (Estimated)

PRIMARY OUTCOMES:
Medical and behavior problems | Through study completion, an average of 5 years
  Collecting medical and behavior health records from individuals affected by Williams syndrome and/or other variants of the chromosome 7q11.23 and analyze potential correlation between genetic factors and physiological, cognitive and behavior manifestations of listed conditions.
Biobank | Through study completion, an average of 5 years
  Collecting biological specimen (saliva, blood, residual tissues) enabling future research.
Quality of life | Through study completion, an average of 5 years
  Making a lost of short-term functional and quality of life outcomes of teens and young adults with WS who are seen through the Armellino Center of Excellence for Williams Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rader, MD, Principal Investigator — University of Pennsylvania; Carolyn Mervis, PhD, Principal Investigator — University of Pennsylvania; Edward Brodkin, MD, Principal Investigator — University of Pennsylvania; Benjamin Yerys, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A limited and de-identified dataset may be available to other researchers
Supporting Information: Study Protocol, ICF
Time Frame: 2027
Access Criteria: Investigators studying Williams syndrome or Dup7 will be welcomed to apply for de-identified limited data set and/or biospecimen. Final decision on sharing will be made by the research committee at the Armellino Center of Excellence.